CLINICAL TRIAL: NCT05323552
Title: Prospective Study Assessing the Laparoscopic Totally ExtraPeritoneal (TEP) Hernia Repair Without Curare and Without Orotracheal Intubation (Free Curare TEP Study).
Brief Title: Hernia Repair Using the Totally ExtraPeritoneal (TEP) Laparoscopic Approach Without Curare and Without Orotracheal Intubation.
Acronym: FREE_CURARE
Status: Recruiting | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: FREE CURARE TEP; 2021-A02830-41 (Other: ANSM)
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Curare

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hernia repair with laparoscopic TEP approach without curare and without orotracheal intubation.: Patients will undergo laparsocopic TEP hernia repair without curare and without orotracheal intubation.
  Interventions: Procedure: Laparoscopic TEP hernia repair without curare and without orotracheal intubation.

INTERVENTIONS:
Procedure: Laparoscopic TEP hernia repair without curare and without orotracheal intubation. — All the techniques and protocols used for this monocentric study are standardized:
  * The anesthesia is general, the anesthetic products administered are identical,
  * ventilation is ensured by the use of a laryngeal mask airway, without curare administered
  * the surgery is an extraperitoneal laparoscopy with an optical trocar under the umbilical and two operators with the placement of a preformed type 3G polypropylene prosthesis
  * the analgesic protocol is free of opioids (Opioid Free Anesthesia - OFA)

SUMMARY:
Laparoscopic treatment of inguinal hernia with the totally extraperitoneal approach (TEP) is indicated for simple and bilateral inguinal hernias. It consists of placing a large prosthesis in the posterior position by direct access to the extra-peritoneal space. This prosthesis is interposed between the defective wall and the peritoneum. Unlike the transperitoneal laparoscopic method, the strictly extraperitoneal approach reduces complications related to contact with the intestinal loops and preserves the peritoneal layer intact.

TEP approach is traditionally performed under general anesthesia with curare and orotracheal intubation.

In the study, we would like to assess this intervention without curare and without standard orotracheal intubation but with a laryngeal mask airway to permit ventilation.

DETAILED DESCRIPTION:
Laparoscopic TEP hernia repair is traditionally performed under general anesthesia with curare and orotracheal intubation. Indeed, according to the French SFAR Recommendations (2018) regarding to curarization and decurarization in anesthesia, it is recommended to administer a curare to facilitate intubation of the trachea. Moreover, the SFAR in these same recommendations specifies that it is probably not recommended to systematically administer curare to facilitate the fitting of a supraglottic airway device (otherwise called a laryngeal mask airway).

The idea of this study is to perform this intervention without curare and without standard orotracheal intubation but with a laryngeal mask airway to permit ventilation. This ventilation technique has already been commonly used by the site for several years. The recent global shortage of curares has led them to increasingly resort to this method during this phase of the global pandemic.

In addition, limiting the patients exposure to curares avoids possible anaphylactic reactions. According to the SFAR, the incidence of anaphylactic reactions to curares varies by country. It was estimated at 184.0 [139.3 - 229.7] in France, 250.9 [189.8 - 312.9] for women and 105.5 [79.7 - 132.0] for men.

The main hypothesis of the study is that the repair of inguinal hernia using the totally extraperitoneal laparoscopic approach (TEP) is feasible without curares and without orotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 or over
2. BMI below 30
3. Non-recurrent unilateral hernia
4. Operating time estimated at less than 60 minutes at the surgeon's discretion
5. Patients eligible to an ambulatory surgical setting at the discretion of the surgeon and the anesthetist
6. Patient informed of the study and agreed to take part.

Exclusion Criteria:

1. Patient under legal protection measures
2. Impossibility of using a laryngeal mask airway
3. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that will undergo a laparoscopic TEP hernia repair without curare and without orotracheal intubation, eligible to an ambulatory surgical setting.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the number of laparoscopic TEP hernia repairs carried out under optimal conditions compared to an intervention requiring adaptation. | During the procedure
  The intervention will be qualified as successful if the following three criteria (i.e. optimal conditions) are validated:
  * No use of curares AND
  * Use of a laryngeal mask airway for the entire duration of the procedure (no use of orotracheal intubation) AND
  * Ambulatory surgical setting, or hospital setting only if not related to the intervention (e.g.: organizational problem of returning home).
  If one of the above criteria is not met, the intervention will be considered as failure for the primary endpoint.

SECONDARY OUTCOMES:
Assessment of the intervention-related ambulatory surgical setting failure. | During the procedure
  Comparison of the proportions of ambulatory surgical settings versus inpatient hospitalizations.
Assessment of the procedure change rate, from a TEP approach to a Trans-Abdominal Pre-Peritoneal approach (TAPP). | During the procedure
  Comparison of the proportions between the TEP approach and the TAPP approach.
Evaluation of the occurrence of post-operative complications during the first month following the intervention. | At 1 month after the procedure
  Collection of Adverse Events until the follow-up visit at 1 month.
Pain assessment | After the procedure and the day after the intervention by phone call
  Pain assessment by a Visual Analogue Scale (VAS) before returning home and then during the phone call the day after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: David Amielh, MD, Principal Investigator — Nouvel Hôpital Privé Les Franciscaines, Nîmes
Locations (1):
- Nouvel Hôpital Privé Les Franciscaines, Nîmes, France

REFERENCES:
- [Background] Fitzgibbons RJ, Richards AT, Quinn TH. Open hernia repair. In: Souba WS, Mitchell P, Fink MP, Jurkovich GJ, Kaiser LR, Pearce WH, et al., editors. ACS surgery: principles and practice. 6th ed. Philadelphia, USA: Decker Publishing Inc.; 2002. p. 828-49.
- [Background] Meyer A, Dulucq JL, Mahajna A. Laparoscopic totally extraperitoneal hernioplasty with nonfixation of three-dimensional mesh: Dulucq's technique. Arq Bras Cir Dig. 2013 Jan-Mar;26(1):59-61. doi: 10.1590/s0102-67202013000100013. English, Portuguese. PMID 23702873
- [Background] Miserez M, Alexandre JH, Campanelli G, Corcione F, Cuccurullo D, Pascual MH, Hoeferlin A, Kingsnorth AN, Mandala V, Palot JP, Schumpelick V, Simmermacher RK, Stoppa R, Flament JB. The European hernia society groin hernia classification: simple and easy to remember. Hernia. 2007 Apr;11(2):113-6. doi: 10.1007/s10029-007-0198-3. Epub 2007 Mar 13. PMID 17353992
- [Background] Baillard C, Bourgain JL, Bouroche G, et al. Actualisations de recommandations - Curarisation et décurarisation en anesthésie. Société Française d'Anesthésie et de Réanimation, 2018.
- [Result] Meyer A, Dulucq JL, Mahajna A. Laparoscopic hernia repair: nonfixation mesh is feasibly? Arq Bras Cir Dig. 2013 Jan-Mar;26(1):27-30. doi: 10.1590/s0102-67202013000100006. English, Portuguese. PMID 23702866
- [Result] Meyer A, Blanc P, Balique JG, Kitamura M, Juan RT, Delacoste F, Atger J. Laparoscopic totally extraperitoneal inguinal hernia repair: twenty-seven serious complications after 4565 consecutive operations. Rev Col Bras Cir. 2013 Jan-Feb;40(1):32-6. doi: 10.1590/s0100-69912013000100006. English, Portuguese. PMID 23538536
- [Result] Dahlstrand U, Sandblom G, Ljungdahl M, Wollert S, Gunnarsson U. TEP under general anesthesia is superior to Lichtenstein under local anesthesia in terms of pain 6 weeks after surgery: results from a randomized clinical trial. Surg Endosc. 2013 Oct;27(10):3632-8. doi: 10.1007/s00464-013-2936-1. Epub 2013 Apr 10. PMID 23572220
- [Result] Neumayer L, Giobbie-Hurder A, Jonasson O, Fitzgibbons R Jr, Dunlop D, Gibbs J, Reda D, Henderson W; Veterans Affairs Cooperative Studies Program 456 Investigators. Open mesh versus laparoscopic mesh repair of inguinal hernia. N Engl J Med. 2004 Apr 29;350(18):1819-27. doi: 10.1056/NEJMoa040093. Epub 2004 Apr 25. PMID 15107485
- [Result] Ozgun H, Kurt MN, Kurt I, Cevikel MH. Comparison of local, spinal, and general anaesthesia for inguinal herniorrhaphy. Eur J Surg. 2002;168(8-9):455-9. doi: 10.1080/110241502321116442. PMID 12549684